CLINICAL TRIAL: NCT00896597
Title: An Open, Randomised Study to Compare the Reproducibility of CTP Rating and NRL972 Pharmacokinetics in Patient Volunteers With Hepatic Cirrhosis.
Brief Title: Reproducibility of Child-Turcotte-Pugh (CTP) Rating and NRL972 Pharmacokinetics in Patients With Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Dr Hans-Jürgen Gruss, Norgine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NRL972-11/2008 (PAIR)
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Hepatic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — NRL972

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NRL972 (Experimental): A single dose of 2 mg NRL972 will be administered on four occasions over a period of up to 6 weeks.
  Interventions: Drug: NRL972

INTERVENTIONS:
Drug: NRL972 — 2 mg NRL972 in 5 mL solution for injection administered as a 15-second intravenous injection on each of four occasions.

SUMMARY:
This is an open, randomized study in patients with different severity stages of hepatic cirrhosis, in which rater pairs will be used for the assessment of the intra- and inter-rater reproducibility of NRL972 pharmacokinetics and CTP sum score. Rating will be performed by 32 to 40 pairs of raters. The raters will perform the required assessments in the capacity of sub-investigators of the phase I (co-ordinating) unit.

Up to 240 patients with clinically established hepatic cirrhosis without confounding end-stage co-morbidity (stable disease) will be studied. Within 30 days of confirmation of eligibility, Visit 1 will take place to determine the investigational parameters (NRL972 pharmacokinetics, clinical laboratory tests, and determination of CTP sum score). At approximate intervals of one week, Visits 2, 3 and 4 will occur, and the investigational parameters will again be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written Informed Consent.
* Gender: male and female (non-childbearing potential = postmenopausal or medically adequate contraception).
* Ethnicity: Any.
* Age: 18 to 80 years of age.
* Patient volunteers with a diagnosis of clinically stable hepatic cirrhosis with a CTP class A, B and C but excluding patient volunteers with the diagnosis of primary biliary cirrhosis, primary sclerosing cholangitis and cystic fibrosis-associated liver disease.
* No previous liver transplantation or intended liver transplantation within the next 6 months after enrollment.
* No previous transjugular intrahepatic portosystemic shunt (TIPS) or portocaval anastomosis (PCA).
* Medically fit to undergo the protocol-defined procedures without undue risk and discomfort.
* No previous participation in a study with an investigational product within 90 days prior to enrolment except epidemiologic or observational studies.

Exclusion Criteria:

* Previous participation in this trial (except for scheduled re-testing in relation to technical difficulties with initial test or rescreening).
* Donation of blood during the last 60 days or a history of excessive blood loss within the last 3 months, assessed using clinical judgement.
* Any donation of germ cells, blood, organs or bone marrow during the course of the study.
* History of any clinically relevant allergy (including hypersensitivity to the IMP).
* Presence of clinical relevant acute or chronic infection (other than chronic viral hepatitis, if applicable).
* Presence of hepatic encephalopathy at grades 3 or 4
* Unstable clinical presentation of hepatic cirrhosis (not allowing completion of participation in the study within 6 weeks).
* Use of confounding concomitant medication (see Section 7.5.7).
* Presence or history of any end-stage (co-)morbidity (excluding the effects of hepatic cirrhosis) such as: malignancy and clinically relevant systemic diseases.
* Presence of primary and/or hepatic malignancy.
* Suspicion or evidence that the patient volunteer is not trustworthy and reliable.
* Suspicion or evidence that the patient volunteer is not able to make a free consent or to understand the information in this regard.
* Primary biliary cirrhosis and primary sclerosing cholangitis.
* Cystic fibrosis.
* Patient volunteers who are employees at the investigational site, relatives or spouses of the investigator.
* Current drug or medication abuse.

Special restrictions for female patient volunteers:

* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation.
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career or lifestyle precludes intercourse with a male partner and women whose partners have been sterilised by vasectomy or other means, unless they meet the following definition of post-menopausal:

  * 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/m or 6 weeks post surgical bilateral oophorectomy with or without hysterectomy or hysterectomy
  * OR are using one or more of the following acceptable methods of contraception:

    * surgical sterilisation (e.g., bilateral tubal ligation, vasectomy)
    * hormonal contraception (implantable, patch, oral), and
    * double-barrier methods (any double combination of: an intrauterine device, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the reproducibility of the CTP sum score with the reproducibility of the pharmacokinetics of NRL972, both assessed by a rater pair, in patients with stable hepatic cirrhosis. | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Gruss, MD, Study Director — Norgine
Locations (1):
- IFE Romania, Timișoara, Romania